CLINICAL TRIAL: NCT07346495
Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of a Single Dose of Remternetug in Healthy Chinese Participants
Brief Title: A Study of Remternetug (LY3372993) in Healthy Chinese Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18470; J1G-GH-LAKE (Other: Eli Lilly and Company)
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Remternetug (Experimental): Remternetug will be administered subcutaneously (SC)
  Interventions: Drug: LY3372993
- Placebo (Placebo Comparator): Placebo will be administered Subcutaneously (SC)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3372993 — Administered SC
  Other Names: Remternetug
  Arms: Remternetug
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The study will evaluate the safety and tolerability of remternetug when given subcutaneously (SC) (under the skin) to healthy Chinese participants. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. The study will last up to 25 weeks, including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, electrocardiogram (ECG), and Magnetic resonance imaging (MRI).
* Participants must be native Chinese. To qualify as Chinese for this study, the participant, the participant's biological parents, and all 4 of the participant's biological grandparents must be of exclusive Chinese descent and born in China.
* Have clinical laboratory test results within normal reference ranges for the population or study site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have a body mass index within the range 18.0 to 28.0 kilograms per square meter (kg/m²), inclusive.
* Are individuals Assigned Male at Birth (AMAB) or individuals Assigned Female at Birth (AFAB) who are individuals not of childbearing potential (INOCBP). Individual of childbearing potential (IOCBP) are excluded from the trial.

Exclusion Criteria:

* Are women who are lactating.
* Have known allergies to remternetug, related compounds, including donanemab, or any components of the formulation.
* Have history of allergies to medications for the emergency treatment of systemic hypersensitivity reactions, including anaphylaxis or infusion reactions (for example, epinephrine, diphenhydramine).
* Have a 12-lead ECG abnormality at screening that, in the opinion of the investigator, increases the risks associated with participating in the study or may confound ECG data analysis.
* Have an abnormal blood pressure or pulse rate as determined by the investigator, or a preexisting history of hypertension.
* Have a history or presence of significant psychiatric disorders.
* Have a brain MRI that demonstrates any clinically significant findings that in the opinion of the investigator may impact the participant's ability to safely participate in the study.
* Have a family history of early onset Alzheimer's disease (AD) (AD diagnosed prior to 65 years of age).
* Have a history or presence of clinically significant multiple or severe drug allergies or severe posttreatment hypersensitivity reactions, including, but not limited to, erythema multiforme major, linear immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis.
* Have history or presence of uncontrolled asthma, significant autoimmune disease, hereditary angioedema, or known history of common variable immune deficiency.
* Have a history or presence of serious or unstable illnesses including cardiovascular, hepatic, renal, gastrointestinal, respiratory, endocrine, psychiatric, immunologic, hematologic disease, or neurological disorders and other conditions that, in the investigator's opinion, could significantly alter the absorption, metabolism, or elimination of drugs; interfere with the analyses in this study; increase risk for study intervention administration; or result in a participant's life expectancy of less than 24 months.
* Have significant neurological disease affecting the central nervous system that may affect the participant's ability to complete the study, including but not limited to dementias, serious infection of the brain, Parkinson's disease, multiple concussions, intracranial hemorrhage, cerebrovascular aneurysm or arteriovenous malformation, or carotid artery occlusion, stroke, unprovoked seizure, epilepsy, or recurrent seizures (except febrile childhood seizures).
* Have donated blood of more than 400 milliliter (mL) within the previous 4 weeks of study screening, or plan for blood donation during the study period.
* Have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Have had significant medical history of dizziness, syncope, or vasovagal attacks within the past 3 years.
* Have used or intend to use over-the-counter, prescription, or Chinese traditional medicines and herbal supplements within 14 days or 5 half-lives (whichever is longer) prior to dosing. Vitamins and mineral supplements not providing more than 100% of the recommended daily amount and thyroid hormone replacement are allowed.
* Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies.
* Have a positive Hepatitis C virus (HCV) antibody test. Participants with a positive HCV antibody test at screening can be included only if a confirmatory HCV ribonucleic acid (RNA) test is negative.
* Show evidence of hepatitis B or positive hepatitis B surface antigen. Other Exclusion Criteria
* Have an average weekly alcohol intake that exceeds 21 units per week for males and 14 units per week for females; 1 unit = 12 ounce (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits.
* Are unwilling to stop alcohol consumption for 48 hours prior to admission to the study site or outpatient visits.
* Smoke more than 10 cigarettes per day or the equivalent including electronic cigarettes, are unwilling to refrain from smoking for approximately 1 hour prior to each ECG and vital sign measurement during the study, or are unable to abide by CRU smoking restrictions.
* Have Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), or Alkaline Phosphatase (ALP) greater than or equal to 1.5× Upper Limit of Normal (ULN) at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through study completion up to 25 weeks

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Remternetug | Day 1 through Day 5
PK: Area Under the Concentration Versus Time Curve (AUC) of Remternetug | Day 1 through Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Xuhui District Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No